CLINICAL TRIAL: NCT05434962
Title: A Non-inferiority Randomized Comparison Between LEFT BUNDLE Branch Area Pacing and Biventricular Pacing for Cardiac Resynchronization Therapy: The LEFT-BUNDLE-CRT Trial
Brief Title: The Left Bundle Cardiac Resynchronization Therapy Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Óscar Cano Pérez (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Sponsor-Investigator, Óscar Cano Pérez, Cardiologist, Spanish Society of Cardiology
Organization: Spanish Society of Cardiology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB-CRT-001
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Left Bundle-Branch Block; Heart Failure; Impaired Left Ventricular Function
Keywords: cardiac resynchronization therapy; conduction ssystem pacing
MeSH Terms: conditions — Bundle-Branch Block; Heart Failure; Ventricular Dysfunction, Left | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac resynchronization therapy (CRT) obtained by stimulating the left branch area (Experimental): The CRT-P/CRT-D device and leads should be implanted according to the physician's standard practice. Only locally approved Medtronic CRT-P/CRT-D generators will be used during the study. It is strongly encouraged the designation of a single and experienced implanting physician at each center for the LBBAP implant procedures.
  During the implant procedure lead impedances, pacing and sensing parameters will be measured using a pacing system analyzer (PSA).
  For LBBAP, the Medtronic 3830 lead will be used. Acceptable LBBAP threshold should be <2,5V@0,5ms.
  Interventions: Device: Cardiac resynchronization therapy
- Cardiac resynchronization therapy (CRT) obtained by biventricular pacing (Active Comparator): The CRT-P/CRT-D device and leads should be implanted according to the physician's manual provided with the devices. Only locally approved Medtronic CRT-P/CRT-D generators will be used during the study.
  Investigators may use any market approved right atrial (RA) pace/sense lead, right ventricular (RV) pacing/defibrillator lead with pace/sense capabilities and any market approved unipolar/bipolar/quadripolar LV pacing lead.
  During the implant procedure lead impedances, pacing and sensing parameters will be measured using a pacing system analyzer (PSA).
  The LV lead should be implanted at a lateral or posterolateral CS branch in a basal or mid ventricular position confirmed by ortogonal fluoroscopic views (RAO and LAO 40º).
  Acceptable LV pacing threshold should be <3V@0,5ms and phrenic nerve stimulation (PNS) margin should be >1V with respect to the pacing threshold
  Interventions: Device: Cardiac resynchronization therapy

INTERVENTIONS:
Device: Cardiac resynchronization therapy — Standard BiV-CRT The CRT-P/CRT-D device and leads should be implanted according to the physician's manual provided with the devices. Only locally approved Medtronic CRT-P/CRT-D generators will be used during the study. The LV lead should be implanted at a lateral or posterolateral CS branch in a basal or mid ventricular position confirmed by ortogonal fluoroscopic views (RAO and LAO 40º). Acceptable LV pacing threshold should be <3V@0,5ms and phrenic nerve stimulation (PNS) margin should be >1V with respect to the pacing threshold.
  LBBAP-CRT The CRT-P/CRT-D device and leads should be implanted according to the physician's standard practice. Only locally approved Medtronic CRT-P/CRT-D generators will be used during the study. During the implant procedure lead impedances, pacing and sensing parameters will be measured using a pacing system analyzer (PSA). For LBBAP, the Medtronic 3830 lead will be used. Acceptable LBBAP threshold should be <2,5V@0,5ms

SUMMARY:
Cardiac resynchronization therapy (CRT) via biventricular (BiV) pacing significantly reduces morbidity and mortality in patients with left bundle branch block (LBBB), impaired LV function and heart failure in spite of optimal medical treatment. CRT positive effects are based on the existence of an electromechanical dyssynchrony induced by the abnormal activation sequence associated with the presence of a left bundle branch block (LBBB), which is thought to be responsible for a negative LV remodeling leading to LVEF impairment and heart failure progression. However, one third of patients undergoing CRT are considered non responders due to different reasons. Recently, left bundle branch area pacing (LBBAP) has emerged as a novel physiological pacing modality aiming for conduction system recruitment in patients with normal or impaired atrioventricular conduction, including patients with LBBB. LBBAP achieves LBBB correction in up to 85% of the cases and thus could be a promising pacing modality for CRT candidates.

DETAILED DESCRIPTION:
Medical device: Only CE-marked CRT-P or CRT-D Medtronic devices locally approved and commercially available (Medtronic 3830 Pacing Lead) shall be used in this protocol.

Indication: Pacing and sensing in the right atrium or ventricle. It is also designed for pacing and sensing in the bundle as an alternative to pacing in the right ventricle in a single or dual chamber pacing system.

Intended use: Patients with an indication for cardiac resynchronization therapy.

Duration of the study: Approximate inclusion period of 18 months

Follow-up: Patients will be followed for 12 months ± 4 weeks after implant

Planned study period: The study is planned to start in Q1 2022

No. of sites: Approximately 11 sites in Spain.

No. of subjects: 176 patients will be enrolled in the study

Study type: Post-market study

Study rationale: Previous studies show 85% implantation success, significant reduction in QRS duration, and significant improvement in NYHA functional class, LVEF, and LV end-diastolic diameter. Left bundle branch pacing could be an alternative to conventional biventricular pacing.

Study design: Multicenter, prospective, randomized, non-inferiority, open.

Objectives of the study:

* Primary objective: The primary objective of the study is to demonstrate that LBBAP is associated with a non-inferior percentage of CRT responders at 6 months follow-up than conventional BiV pacing using a conventional CS lead in patients with CRT indications according to current guidelines. Positive CRT response will be defined either by an improved Clinical Composite Score or ≥15% reduction in left ventricular end-systolic volume at 6 months follow-up
* Secondary objectives: To evaluate reverse ventricular remodeling response and dyssynchrony parameters based on echocardiographic data at 6 and 12 months follow-up. To asess clinical outcome using the Clinical Composite Score, 6 minute walking test, quality of life measurements (EuroQuol EQ 5-D) at 6 and 12 months follow-up. To evaluate HF related hospitalizations at 6 and 12 months follow-up. To evaluate mortality (global and cardiovascular) and need for cardiac transplantation at 6 and 12 month follow-up. To evaluate incidence of ventricular arrhythmias at 6 and 12 month follow-up. To evaluate differences in CRT response depending on the final LBBAP modality (LBBP vs deep septal pacing). To evaluate device related complications at 6 and 12 month follow-up.

Primary Outcome Measures: Improved Clinical Composite Score or ≥15% reduction in left ventricular end-systolic volume at 6 months follow-up.

Participating sites:

* Hospital Universitario y Politécnico La Fe, Valencia
* Hospital Clinic de Barcelona
* Hospital Virgen de las Nieves, Granada
* Hospital Virgen de la Arrixaca, Murcia
* Hospital Puerta de Hierro, Madrid
* Hospital General de Alicante
* Hospital Bellvitge, Barcelona
* Hospital 12 de Octubre, Madrid
* Hospital Universitario Lozano Blesa, Zaragoza
* Hospital Juan Ramón Jiménez, Huelva
* Hospital Universitario San Cecilio, Granada

Study population: Subjects 18 years of age or older will be included in the study. Both sexes are eligible to participate. Subjects must present a left bundle branch block (according to Strauss criteria) with indication of CRT class I or IIa according to clinical practice guidelines. A selection of the subjects will be made before inclusion following the selection clinical investigation plan. After confirming that the subject meets the inclusion criteria and does not meet the exclusion criteria, they will be included in the clinical study.

Study population criteria:

* Inclusion criteria: age > 18 years; Class I or IIa indication for CRT according to current ESC or ACC/AHA/HRS guidelines; left bundle branch block according to Strauss criteria; Signed and dated informed consent.
* Exclusion criteria: Pregnant woman; Permanent or long-lasting atrial fibrillation; Previous CRT device; Previous PM/ICD with ventricular pacing > 10%; Conventional pacemaker indication; Nonspecific IVCD (intraventricular conduction delay); Unstable angina, acute Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG), Percutaneous Coronary Angioplasty (PCI), valve repair or replacement within 90 days prior enrollment; Indication for valve repair or replacement; Already included in another clinical study that could confoud the results of the present study; Life expectancy < 12 months.

Device Implantation Procedure: CRT obtained by biventricular pacing vs. CRT obtained by stimulating the left branch area.

Follow-up: Follow-up should be carried out with pre-established periodic clinical appointments 3, 6, and 12 months after hospital discharge. In the follow-up, routine examinations such as vital signs, electrocardiogram and echocardiogram (6 and 12 months) are recorded to check the evaluation of the reverse ventricular remodeling response and asynchrony parameters based on echocardiographic data.

Statistical considerations: Once patients have signed the informed consent at baseline visit, patients will be considered as "Enrolled population" in the statistical analysis. The sample size is based on the primary endpoint: Improved Clinical Composite Score or ≥15% reduction in left ventricular end-systolic volume at 6 months follow-up, showing that LBBAP is non-inferior to BiV-CRT. Accounting for a global attrition rate of 10% and considering the block size for randomization, 176 patients shall be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Class I or IIa indication for CRT according to current ESC or ACC/AHA/HRS guidelines
* left bundle branch block according to Strauss criteria
* Signed and dated informed consent

Exclusion Criteria:

* Pregnant woman
* Permanent or long-lasting atrial fibrillation
* Previous CRT device
* Previous PM/ICD with ventricular pacing > 10%
* Conventional pacemaker indication
* Nonspecific IVCD (intraventricular conduction delay)
* Unstable angina, acute Myocardial Infarction (MI), Coronary Artery Bypass Graft (CABG), Percutaneous Coronary Angioplasty (PCI), valve repair or replacement within 90 days prior enrollment
* Indication for valve repair or replacement
* Already included in another clinical study that could confoud the results of the present study
* Life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
CRT response | 6 months follow-up
  Positive CRT response will be defined either by an improved Clinical Composite Score or ≥15% reduction in left ventricular end-systolic volume

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 6 and 12 months follow-up
  To evaluate left ventricular ejection fraction at 6 and 12 months follow-up
Clinical outcome | 6 and 12 months follow-up
  Assessed by the Clinical Composite Score
Exercise capacity | 6 and 12 months follow-up
  Assessed by 6 minute walking test
The EQ-5D three-level version (EQ-5D-3L) | 6 and 12 months follow-up
  Is a generic measure of health status consisting of 2 parts. The first assesses health in five dimensions (mobility, selfcare, usual activities, pain / discomfort, anxiety / depression), each of which has 3 levels of response (no problems, some problems, extreme problems / unable to). This part of the questionnaire provides a descriptive profile that can be used to generate a health state profile. Each health state can potentially be assigned a summary index score based on societal preference weights for the health state. Health state index scores generally range from less than 0 (where 0 is a health state equivalent to death; negative values are valued as worse than death) to 1 (perfect health), with higher scores indicating higher health utility. The second part consists of a VAS on which the patient rates his / her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health)
Heart Failure Hospitalizations | 6 and 12 months follow-up
  Assessment of heart failure hospitalizations
Mortality | 6 and 12 months follow-up
  To evaluate mortality (global and cardiovascular)
Cardiac transplantation | 6 and 12 months follow-up
  To evaluate the need for cardiac transplantation during follow-up
Ventricular arrhythmias | 6 and 12 month follow-up
  To evaluate incidence of ventricular arrhythmias (clinical and registered by the ICD/PM)
Device related complications | 6 and 12 month follow-up
  Device related complications needing re-intervention

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital General Universitario de Alicante Doctor Balmis, Alicante, Alicante
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Universitario San Cecilio, Granada, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva, Huelva
  - Hospital 12 Octubre, Madrid, Madrid
  - Hospital Universitario Puerta De Hierro, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: No